CLINICAL TRIAL: NCT05376787
Title: The Purpose of This Study is to Verify the Performance of the Neutral Electrode (NE) Adhesives in Accordance With the Testing Specified in IEC 60601-2-2:2017, Section 201.15.101.7, Pull Test.
Brief Title: Verify the Performance of the Neutral Electrode (NE) Adhesives
Status: Completed | Type: Observational
Sponsor: Medline Industries (Industry)
Collaborators: F2 Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: F2P27778
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: Adhesion of the Neutral Electrode 21pad

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy Subjects: Participants must be willing to comply with all study procedures Participants must be willing to shave, or to have shaved, the sites where the neutral electrodes will be placed.
  Interventions: Device: Medline NE Grounding Pad

INTERVENTIONS:
Device: Medline NE Grounding Pad — Split Universal Grounding Pads

SUMMARY:
The purpose of this research study is to determine the neutral electrode 21pad adhesion to the skin in accordance with international standard IEC 60601-2-2 section 201.15.101.7. A neutral electrode is placed on the body of patients undergoing surgery that involves the use of electric current, to protect them from the harmful effects of the electricity.

DETAILED DESCRIPTION:
Two neutral electrodes will be applied to the front of your thighs. The study staff will set up and attach a pulley system to the neutral electrodes. The purpose of the pulley system is to apply a force pulling the neutral electrode away from your body. The force will be applied for 10 minutes on each neutral electrode in one direction, and then for another 10 minutes in a second direction. Site staff will mark any areas of separation and the neutral electrodes will be removed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be willing to comply with all study procedures
* Participants must be willing to shave, or to have shaved, the sites where the neutral electrodes will be placed.

Exclusion Criteria:

* The participant has any skin conditions (e.g. eczema, sensitivities, allergies to adhesives, sunburn, etc.) at the application sites that might be adversely affected by the application of an adhesive pad.
* The participant is pregnant or breastfeeding.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of at least 10 males and 10 females. Participants must be healthy and of at least 18 years of age. Participants must also fit inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- F2 Labs, Damascus, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Subjects: Subjects must be 18 years old or over, willing to shave or have shaved the sites where the neutral electrodes will be placed. Subjects also must not be pregnant, breastfeeding, have skin conditions (such as eczema, sensitivities, allergies to adhesives, sunburn).
  Medline NE Grounding Pad: Split Universal Grounding Pads
Period: Overall Study
Arm/Group | Healthy Subjects
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Tests With No More Than 5% Separation - Neutral Electrode (NE) Adhesive Separation
Description: To determine the percentage of adhesion separation by only measuring test results that had no more than 5% of the NE adhesive area separated.
  At Point A where the NE connects to the pad, connect a cord to pull on the cable. Pull for 10 to 10.25 minutes, in a plane parallel to the NE pad and in a direction away from the center of the pad, with 10 to 11N (1.02 to 1.12kg) of force in the direction along the minor dimension of the pad. Set the height of the pulley so that the direction of pull shall be approximately co-planer with the plane of the connection point of the NE. The pull shall be performed by a cord connected to the NE at the cable connection point. See Figure 2 for the pull set up. The weights provide the required pull force. Start timer. At 10 mins, change direction of pull to y direction by rotating the pulley system 90 degrees as shown in Figure 2 - apply 10 to 11 N force at Point A in direction of y ray which is in a plane parallel to the pad.
  Start timer. At 10 mins
Time Frame: Up to 20 minutes - (10 minutes w. Pull for 10 to 10.25 minutes, in a plane parallel to the NE pad & At 10 mins, change direction of pull to y direction)
Population: Healthy participants. Adhesion testing was done on each leg, so there was a total of two tests per participant. A total of 40 tests were done.
Measure: Number; unit: Tests
Units Other Than Participants: Test legs
Arm/Group | Healthy Subjects
Number analyzed (Participants) | 20
Number analyzed (Test legs) | 40
Tests | 39

ADVERSE EVENTS:
Time Frame: Up to 20 minutes
Arm/Group | Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT05376787/Prot_SAP_000.pdf